CLINICAL TRIAL: NCT00605813
Title: Special Investigation Of Long Term Use Of J ZOLOFT.
Brief Title: Special Investigation Of Long Term Use Of Sertraline.
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0501091
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2012-09-10 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Depression; Panic Disorder
MeSH Terms: conditions — Depression; Panic Disorder | interventions — Sertraline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sertraline hydrochloride.: Patients taking Sertraline hydrochloride.
  Interventions: Drug: Sertraline hydrochloride

INTERVENTIONS:
Drug: Sertraline hydrochloride — J ZOLOFT® Tablets 25 mg and J ZOLOFT® Tablets 50 mg. J ZOLOFT is Brand name in Japan.
  Dosage, Frequency: According to Japanese LPD, "The usual initial dose of J ZOLOFT in adults is 25 mg daily as sertraline and then gradually increased up to 100 mg, which should be given orally once daily. The dose may be adjusted within the range not exceeding 100mg according to the patient's age and symptoms".
  Duration: According to the protocol of A0501091, the duration of the investigation for findings regarding safety and efficacy of a patient is from the first drug administration to the 52 weeks after the first administration.
  Other Names: J Zoloft, Zoloft

SUMMARY:
Special investigation of long term use of sertraline, 52 Week Observation, Long-Term Safety. The objective of this "Special investigation" is to collect information about 1) adverse drug reactions not expected from the LPD (unknown adverse drug reactions), 2) the incidence of adverse drug reactions in this surveillance, and 3) factors considered to affect the safety and/or efficacy of this drug regarding long time use.

DETAILED DESCRIPTION:
All the patients for whom an investigator prescribes the first sertraline hydrochloride should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

The patients who take sertraline hydrochloride for longer than the duration of 16 weeks among the patients enrolled in A0501090 (Drug Use Investigation of J Zoloft).

Exclusion Criteria:

Patients not taking sertraline hydrochloride.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients to whom an investigator involved in A0501091 prescribes sertraline hydrochloride.
Sampling Method: Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline: Participants taking Sertraline according to Japanese Package Insert
Period: Overall Study
Arm/Group | Sertraline
Started | 542
Completed | 517
Not Completed | 25
Not completed — Protocol Violation | 25

BASELINE CHARACTERISTICS:
Arm/Group | Sertraline
Number analyzed (Participants) | 517
Age, Customized [Number; unit: participants]
  <65 years | 447
  >=65 years | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 311
  Male | 206
Target Disease [Number; unit: participants] — The target disease which was diagnosed by investigator
  participants
    Depression/Depressed State | 426
    Panic Disorder | 44
    Depression/Depressed State and Panic Disorder | 21
    Other than those Above | 26
Target Disease Severity [Number; unit: participants] — The severity of target disease which was diagnosed by investigator
  participants
    Mild | 111
    Moderate | 362
    Severe | 44
Complications [Number; unit: participants] — Complications is the patient's current experiences with illnesses, operations, injuries and treatments. The physician of this survey made the diagnosis. (e.g. hypertension, diabetes, etc.)
  participants
    Present | 198
    Absent | 319
Concomitant Drug [Number; unit: participants] — Concomitant drugs is the drugs which participant had taken during the observation period of this study to treat for participant's illnesses, injuries etc. The physician of this survey listed all of concomitant drugs. (e.g. paroxetine, milnacipran, etc.)
  participants
    Present | 470
    Absent | 47
Starting Dose [Number; unit: participants] — Starting dose of each participant enrolled in this study
  participants
    25 mg | 348
    50 mg | 144
    75 mg | 10
    100 mg | 6
    Other than those Above | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Related Adverse Events (TRAEs) Not Expected From Japanese Package Insert
Time Frame: Baseline up to 52 weeks
Population: The safety analysis population consists of the cases that satisfy the participants conditions and in whom administration of Sertraline was confirmed.
Measure: Number; unit: events
Groups:
- Sertraline Hydrochloride: Participants who took Sertraline according to Japanese Package Insert
Arm/Group | Sertraline Hydrochloride
Number analyzed (Participants) | 517
events
  Erectile dysfunction | 2
  Dissociative disorder | 1
  Completed suicide | 1

2. Primary Outcome: Number of Participants of Treatment Related Adverse Events (TRAEs)
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Definition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product.
Time Frame: Baseline up to 52 weeks
Population: Safety analysis population included all enrolled subjects who had received at least 1 confirmed, administration of Sertraline.
Measure: Number; unit: events
Groups:
- Sertraline: Participants who took Sertraline according to Japanese Package Insert
Arm/Group | Sertraline
Number analyzed (Participants) | 517
events | 44

3. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Renal Dysfunction
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertralinedine to determine whether with or without renal dysfunction is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Without Renal Dysfunction: Participants without renal dysfunction who took Sertraline according to Japanese Package Insert
- With Renal Dysfunction: Participants with renal dysfunction who took Sertraline according to Japanese Package Insert
Arm/Group | Without Renal Dysfunction | With Renal Dysfunction
Number analyzed (Participants) | 513 | 4
participants | 42 | 2
Statistical Analysis 1: Comparison: Without Renal Dysfunction vs With Renal Dysfunction; The risk factor tested was "renal dysfunction". The null hypothesis is there is no difference between "with and without renal dysfunction" in the participants of responders; Test type: Superiority or Other; p = 0.003, Chi-squared — not adjusted, p=0.050

4. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Past Medical History of Other Illness
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertralinedine to determine whether with or without past medical history of other illness is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Without Past Medical History of Other Illness: Participants without past medical history of other illness who took Sertraline according to Japanese Package Insert
- With Past Medical History of Other Illness: Participants with past medical history of other illness who took Sertraline according to Japanese Package Insert
Arm/Group | Without Past Medical History of Other Illness | With Past Medical History of Other Illness
Number analyzed (Participants) | 436 | 81
participants | 28 | 16
Statistical Analysis 1: Comparison: Without Past Medical History of Other Illness vs With Past Medical History of Other Illness; The risk factor tested was "past medical history of other illness". The null hypothesis is there is no difference between "with and without past medical history of other illness" in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

5. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Non-Pharmaceutical Therapies
Description: Number of participants with responders of Sertraline to determine whether with or without non-pharmaceutical therapies is significant factor
Time Frame: Baseline up to 52 weeks
Population: The efficacy analysis population consists of the evaluable cases in accordance with the analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Groups:
- With Non-pharmaceutical Therapies: Participants with non-pharmaceutical therapies who took Sertraline according to Japanese Package Insert
- Without Non-pharmaceutical Therapies: Participants without non-pharmaceutical therapies who took Sertraline according to Japanese Package Insert
Arm/Group | With Non-pharmaceutical Therapies | Without Non-pharmaceutical Therapies
Number analyzed (Participants) | 155 | 266
participants | 141 | 255
Statistical Analysis 1: Comparison: With Non-pharmaceutical Therapies vs Without Non-pharmaceutical Therapies; The risk factor tested was "non-pharmaceutical therapies". The null hypothesis is there is no difference between "with or without non-pharmaceutical therapies" in the participants of responders; Test type: Superiority or Other; p = 0.040, Chi-squared — not adjusted, p=0.050

6. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Present or Past History of Intentional Suicidal Ideation (Including Suicide Attempt)
Description: Number of participants with responders of Sertraline to determine whether present or past history of intentional suicidal ideation (including suicide attempt) is significant factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Past History of Intentional Suicidal Ideation: Participants with past history of intentional suicidal ideation (including suicide attempt) who took Sertraline according to Japanese Package Insert
- Present History of Intentional Suicidal Ideation: Participants with present intentional suicidal ideation (including suicide attempt) who took Sertraline according to Japanese Package Insert
Arm/Group | Past History of Intentional Suicidal Ideation | Present History of Intentional Suicidal Ideation
Number analyzed (Participants) | 35 | 64
participants | 29 | 63
Statistical Analysis 1: Comparison: Past History of Intentional Suicidal Ideation vs Present History of Intentional Suicidal Ideation; The risk factor tested was "present or past history of intentional suicidal ideation". The null hypothesis is there is no difference between "present or past history of intentional suicidal ideation (including suicide attempt)" in the participants of responders; Test type: Superiority or Other; p = 0.004, Chi-squared — not adjusted, p=0.050

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sertraline
Serious Adverse Events (participants affected / at risk) | 2/517
Other Adverse Events (participants affected / at risk) | 44/517
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=517)
Dissociative disorder (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=517)
Somnolence (Nervous system disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 7 (7)
Mania (Psychiatric disorders) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Ejaculation delayed (Reproductive system and breast disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Dissociative disorder (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Weight increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.